CLINICAL TRIAL: NCT06864884
Title: A Phase 1 Randomized, Placebo-Controlled, Blinded Study Evaluating the Safety, Tolerability, and Pharmacokinetics of ARC-001 in Participants Undergoing Third Molar Extraction
Brief Title: A Phase 1 Study of ARC-001 in Participants Undergoing Third Molar Extraction
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arcato Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARC-001-101
Record Dates: First submitted 2025-02-26; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Post Operative Pain; Third Molar Extraction Surgery
Keywords: wisdom teeth surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARC-001 (Experimental): 0.75 mL gel emulsion with active ingredient applied once to the surgical site.
  Interventions: Drug: ARC-001
- Placebo (Placebo Comparator): 0.75 mL gel without active ingredient applied once to the surgical site.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: ARC-001 — Gel formulation containing investigational anesthetic.
  Arms: ARC-001
Drug: Placebo gel — Gel that contains no active ingredients.
  Arms: Placebo

SUMMARY:
The study will test the investigational product gel against placebo (which contains no active ingredient) to determine if it is safe after wisdom tooth extraction. The main questions the study will answer are:

1. How much of the investigational product is absorbed in the blood?
2. Are there side effects?

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* In generally good health
* BMI 18 to 38kg/m²
* Scheduled to undergo wisdom teeth extraction

Exclusion Criteria:

* Serious medical condition
* Clinically significant abnormal lab values
* Blood donation in the last 60 days, or plasma donation in the last 7 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 28 Days
  To evaluate the safety and tolerability of ARC-001 Gel compared to placebo by comparing the incidence of oral treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) through oral exam for soft tissue health using the modified Landry Index and evaluation of the presence or absence of dry socket.

CONTACTS AND LOCATIONS:
Locations (1):
- CenExel JBR, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No